CLINICAL TRIAL: NCT03826810
Title: Effect of Low-intensity Laser and Photodynamic Therapy on Infected Dentin of Permanent Teeth With MIH - Controlled Clinical Trial
Brief Title: Effect of Low-intensity Laser and Photodynamic Therapy on Infected Dentin of Permanent Teeth With MIH
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Leticia
Record Dates: First submitted 2019-01-29; First posted 2019-02-01 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-01

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical evaluations of complete removal of caries lesion, microbiological and radiographic analysis were made by two blind examiners, who did not know to which group the participants belonged.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aPDT + ART group (Experimental): In this group, both aPDT and ART were performed.
  Interventions: Radiation: aPDT; Procedure: ART
- ART group (Experimental): In this group, only ART was performed.
  Interventions: Procedure: ART

INTERVENTIONS:
Radiation: aPDT — For the aPDT the PapacarieMblue (Fórmula e Ação) was used. It was left for 5 minutes in the cavity. The carious tissue was removed and the application of the PapacarieMblue was repeated. The tissue was then irradiated in a single spot with a red laser, of wavelength of 660 nm, for 300 s, with the energy of 500mJ. These parameters were also applied in the vestibular root of the teeth, to try and prevent sensitivity.
  Arms: aPDT + ART group
Procedure: ART — Removal of infected dentin with a curette only, followed by cavity cleaning and restoration with glass ionomer cement.

SUMMARY:
The objective of this research was to evaluate the clinical effect of photodynamic therapy on dentin infected by caries lesion in permanent teeth with Molar Incisor Hypomineralization (MIH). The study was composed of Groups (1 and 2). The methodology was based on the selection of patients from 6 to 12 years of age with permanent molar teeth, randomly divided. The selected teeth had deep dentin caries lesions on the occlusal surface, and sensitivity, indicated for clinical restorative treatment. Photodynamic therapy was applied with the use of low-intensity laser in permanent teeth selected for the treatment of infected dentin in G1. In this group, antimicrobial photodynamic therapy (aPDT) and atraumatic restorative treatment (ART) were made. In G2, only ART was performed. The teeth were restored with high viscosity glass ionomer cement. All patients had clinical and radiographic follow-up with a time interval of 6 and 12 months. Data were submitted to descriptive statistical analysis. For the evaluation of the association of categorical variables like age and gender, the Chi-square test and Fisher's exact test were used. To analyze the correlation between the continuous variables, the Pearson correlation test was applied. ANOVA and Kruskal-Wallis were applied for the analysis of dentin density in the radiographic images scanned and the microbiological results for colony forming units.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children, without systemic alterations;
* Collaborative children;
* Present at least one permanent molar with active and acute caries lesion in dentin, not exceeding 2/3 and involving only the occlusal, with direct vision and access, without clinical and radiographic signs and symptoms of pulp involvement.

Exclusion Criteria:

* Child with systemic impairment;
* Non-cooperative behavior;
* Carious lesion of Class II, III, IV or V type of Black;
* Clinically: carious lesion involving enamel, deficient restorations, small carious lesions in dentin (without access to hand excavators), occult caries lesions, clinical sign and/or symptom of pulp involvement, clinical impossibility of restoration;
* Radiographically: evidence of pulpal involvement, carious lesion extending beyond 2/3 of the dentin.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change in dentin sensitivity | Before and immediately after treatment.
  Prior to removal of carious tissue, the volunteers responded to the Visual Analogue Scale (VAS), following this protocol: gauze isolation of neighboring teeth and air jet in the tooth with MIH for 3 to 5 seconds. The evaluation of the sensitivity through the VAS was repeated at the end of the procedure, after Atraumatic Restorative Treatment (ART).

SECONDARY OUTCOMES:
Change in colony forming units | Before and immediately after treatment.
  Microbiological specimens were collected from the surface of the dentin before and immediately after the treatment, for later counting of colony forming units.
Change in dentin density | After 6 and 12 months.
  The objective was to quantitatively determine the gray tones of the affected dentin region just below the glass ionomer restoration, whose radiographic control for visualization of the healthy dentin allows the clinical evaluator of the study to compare the treated groups with the density of the remaining dentin in discussion. The statistical analysis of the optical density were made according to the mixed effects model.
Change in the presence of cavity filling | After 6 and 12 months.
  The evaluation scores will be evaluated based on the results of studies by other authors (Frencken, et al., 1996). Digital photos (Canon Sx500 IS Camera) will be taken of all the teeth and, from these photographs, the teeth will be classified as follows:
  0 = present, without defect.
  1. = present, small defects in the margin less than 0.5 mm deep, no need for repair.
  2. = present, small defects in the margin of 0.5 to 1 mm depth, needs repair.
  3. = present, gross defects in the margin of 1 mm or more in depth, needs repair.
  4. = absent, restoration almost / completely lost, needs treatment.
  5. = absent, other treatment was performed for any other reason.
  6. = tooth missing due to any reason.
  7. = present, surface wear less than 0.5 mm, no need for replacement.
  8. = present, surface wear greater than 0.5 mm, need replacement.
  9. = impossible to diagnose.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdades Integradas Da União Educacional Do Planalto Central, Gama, Federal District, Brazil